CLINICAL TRIAL: NCT03802032
Title: Effect of Topical Xylocaine for Pain Relief During Hysterosalpingography Among Infertile Women in Zaria, Nigeria: A Randomised Controlled Trial.
Brief Title: Topical Analgesia for Pain Relief in Hysterosalpingography
Acronym: HSG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahmadu Bello University Teaching Hospital (Other)
Responsible Party: Principal Investigator, Anisah Yahya, Doctor, Ahmadu Bello University Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ahmadu Bello University
Record Dates: First submitted 2019-01-10; First posted 2019-01-14 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Infertility, Female
Keywords: infertility; hysterosalpingography; pain
MeSH Terms: conditions — Infertility, Female; Infertility; Pain | interventions — K-Y jelly

STUDY DESIGN:
Intervention Model Description: A randomised controlled trial
Who Masked: Care Provider
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): 15g of Topical Xylocaine gel
  Interventions: Drug: Lidocaine Gel
- Control group (Placebo Comparator): 15g of KY Jelly
  Interventions: Drug: KY jelly

INTERVENTIONS:
Drug: Lidocaine Gel — topical lidocaine gel
  Arms: Study Group
Drug: KY jelly — topical KY jelly
  Arms: Control group

SUMMARY:
The study will involve giving topical analgesia or placebo and then assessing pain and satisfaction during and after the procedure in order to see wed to the placebo.hether the topical analgesia has helped in decreasing pain associated with the procedure and also whether it has increasedd satisfaction with the procedure compar

DETAILED DESCRIPTION:
STUDY DESIGN:

The study will be a double blind randomized controlled trial. Group A:The study group will be given topical Xylocaine (2% Lidocaine) before the procedure.

Group B:The control group will be given topical K-Y jelly (water based lubricant) before the procedure.

The participants and the radiologist will be blinded at the point of drug administration.

SAMPLE SIZE DETERMINATION:

The formula below was used to calculate the sample size n= (Zα + Zβ)2S2 d2

Assuming a difference in mean pain score among groups of 1.5 and using a standard deviation of of 3.15.

Zα = standard normal deviate. Zβ = power = 95% = 1.64. S = standard deviation = 3.1. D = mean difference in pain score = 1.5 n = (1.96 + 1.64)2 x 3.12 1.52

n = 55 Sample size per group will be rounded up to 60

SAMPLING APPROACH:

A probability sampling method will be used. Simple random sampling using a computer generated table of random numbers will be used. The WINPEPI version 11.65 software will generate the table of random numbers. The numbers 001-140 will be randomly allocated to two groups A and B. Group A will be the study group and group B will be the control group (see appendix). Each number from the table of random numbers will be copied on separate paper and then sealed in a brown envelope. The envelopes will then be kept inside a box after shuffling.

Each patient will be allocated to the group that the number she picks corresponds to on the computer printout. The numbers were made up to 140 to make up for patients that may eventually drop out from the study.

.

SAMPLING RECRUITEMENT:

Women that fulfil the inclusion criteria will be recruited from radiology department as they present for Hysterosalpingogram. After obtaining a written consent, participants will be requested to pick one of the brown envelopes which will contain the randomization group.

BLINDING The drugs to be used (K-Y Jelly and Xylocaine gel) are identical.

DATA COLLECTION METHOD:

An informed written consent will be obtained from participants. Psychological support will be given to the participant by a nurse after the procedure has been explained to the participant. A questionnaire will then be filled. The participant will then be requested to pick an envelope that represents the study number. A detailed explanation about the VAS and its application was given personally to each woman before the procedure. An interviewer administered questionnaire will be used to obtain information on socio-demographic characteristics, reproductive profile, previous history of the procedure and experience with analgesia.

The analgesic or placebo will be applied to the cervix (15ml) using a vaginal applicator 10 minutes before the procedure.

The procedure will then be done using standard clinical protocol. The pain rating scale will be used to evaluate pain during from zero (no pain) to ten (worst possible pain) will be explained to the client. The visual scale comparison to happy, glum, sad and horrified faces will also be explained to the patient.

Pain assessment will be done during the procedure at the following steps:

1. After application of speculum.
2. After cervical manipulation (application of tenaculum and catheter).
3. After filling the uterus with contrast medium.
4. After withdrawal of speculum and catheter.
5. Thirty minutes after completing the procedure.

The Likert scale will be used to assess patient satisfaction following pain management.

.

ELIGIBILITY:
Inclusion Criteria:

* All women that are sent in to the department of radiology for Hysterosalpingogram as part of evaluation for infertility that give consent.

Exclusion Criteria:

* Women that present for hysterosalpingography for other indications apart from infertility and those that have history of allergy to xylocaine and/or K-Y jelly.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — based on biological gender
Enrollment: 120 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-12-22 (Actual); Study Completion 2019-12-22 (Actual)

PRIMARY OUTCOMES:
Pain perception | witthin 45 minutes of the procedure
  The pain score based on visual pain scale that assesses pain perception. It is a scale of 0 to 10.
  0 = absence of pain.
  1. = discomfort
  2. = mild pain.
  3. = annoying pain.
  4. = nagging pain.
  5. = distressing pain.
  6. = miserable.
  7. = intense
  8. = Dreadful.
  9. = worse possible
  10. = unbearable

SECONDARY OUTCOMES:
Patients Satisfaction with procedure | witthin 45 minutes of the procedure
  Satisfaction with the procedure based on Likert scale. The scale is from 1 to 5.
  1. = Very dissatisfied.
  2. = Dissatisfied..
  3. = Neither satisfied nor dissatisfied.
  4. = Satisfied.
  5. = Very satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Anisah Yahya, MBBS, Principal Investigator — Ahmadu Bello University Zaria
Locations (1):
- Ahmadu Bello University Teaching Hospital Shika-Zaria, Zaria, Kaduna State, Nigeria

IPD SHARING:
Plan to Share IPD: Yes
obtained data and result will be shared
Supporting Information: Study Protocol, CSR
Time Frame: within 6 months of completion
Access Criteria: free